CLINICAL TRIAL: NCT00358020
Title: A Phase II, Multi-Center, Open Label Study Of Melphalan, Prednisone, Thalidomide And Bortezomib In Advanced And Refractory Multiple Myeloma Patients
Brief Title: Melphalan, Prednisone, Thalidomide And Bortezomib In Advanced And Refractory Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05141; MPTV
Record Dates: First submitted 2006-07-27; First posted 2006-07-28 (Estimated); Last update posted 2006-12-04 (Estimated); Status verified 2006-11

CONDITIONS: Multiple Myeloma
Keywords: MYELOMA, THALIDOMIDE, BORTEZOMIB
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Thalidomide; Bortezomib

INTERVENTIONS:
Drug: THALIDOMIDE
Drug: BORTEZOMIB

SUMMARY:
The purpose of this study is to evaluate the safety and the efficacy of the association of Melphalan/Prednisone/Thalidomide/VELCADE (MPTV) as salvage treatment in advanced and refractory myeloma patients. This association might further increase the response rate achieved by the standard oral MP regimen.

DETAILED DESCRIPTION:
In Multiple Myeloma (MM) patients, the conventional treatment is the oral combination melphalan and prednisone (MP). thalidomide has been widely used in myeloma, it has been proved clinical effective in refractory myeloma patients, it acts sinergistically in association with dexamethasone. In newly diagnosed patients, the combination oral MP plus thalidomide increased the partial and complete response rate.Bortezomib represents a novel class of anti-cancer drugs, it is active in patient with multiple myeloma who are refractory to conventional chemotherapy. In a preliminary report, the combination of VELCADE and Thalidomide induced a remarkable 60% PR rate in advanced refractory myeloma patients. This study will evaluate the safety and the efficacy of the association of Melphalan/ Prednisone/Thalidomide/VELCADE (MPTV) as salvage treatment in advanced and refractory myeloma patients. This association might further increase the response rate achieved by the standard oral MP regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient is of a legally consenting age as defined by local regulations.
* Patient is, in the investigator(s) opinion willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
* Male patient agrees to use an acceptable method for contraception (i.e., condom or abstinence) for the duration of the study.
* Patient was previously diagnosed with multiple myeloma based on standard criteria.
* Patient is relapsed or refractory after one or two lines of treatment including high-dose chemotherapy with stem cell support, conventional poli-chemotherapy, thalidomide- and melphalan-based regimens.
* Patient has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, greater than 1 g/dL of IgG M-Protein and greater than 0.5 g/dL of IgA M-Protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours.
* Patient has a Karnofsky performance status ≥60%.
* Patient has a life-expectancy >3 months.
* Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1, before study drug administration):
* Platelet count ≥75 x 109/L without transfusion support within 7 days before the test.
* Absolute neutrophil count (ANC) ≥ 0.75 x 109/L without the use of growth factors.
* Corrected serum calcium ≤14 mg/dL (3.5 mmol/L).
* Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal (ULN).
* Alanine transaminase (AST): ≤ 2.5 x the ULN.
* Total bilirubin: ≤ 1.5 x the ULN.
* Calculated or measured creatinine clearance: ≥20 mL/minute.

Exclusion Criteria:

* Patient has an absolute neutrophil count <0.75 × 109/L within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance <20 mL/minute within 14 days before enrollment.
* Patient has ≥Grade 2 peripheral neuropathy within 14 days before enrollment.
* Patient has known hypersensitivity to bortezomib, boron, mannitol or thalidomide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-11; Study Completion 2008-12

PRIMARY OUTCOMES:
SAFETY AND EFFICACY

SECONDARY OUTCOMES:
PROGRESSION FREE SURVIVAL AND OVERALL SURVIVAL

CONTACTS AND LOCATIONS:
Overall Officials: MARIO BOCCADORO, MD, Principal Investigator — DIVISIONE DI EMATOLOGIA DELL'UNIVERSITA' DI TORINO, AZIENDA OSPEDALIERA SAN GIOVANNI BATTISTA, TORINO, ITALY; ANTONIO PALUMBO, MD, Study Director — DIVISONE DI MEATOLOGIA DELL'UNIVERSITA' DI TORINO, AZIENDA OSPEDALIERA SAN GIOVANNI BATTISTA, TORINO, ITALY
Locations (7):
- Italy (7):
  - Divisione Di Ematologia, Ospedale Centrale, Bolzano, BOLZANO
  - Unità Operativa Complessa Di Ematologia, Presidio Ospedaliero Dell'Annunziata, Azienda Ospedaliera Di Cosenza, Cosenza, COSENZA
  - Divisione Di Ematologia E Trapianto Di Midollo Osseo, Azienda Ospedaliera Cervello, Palermo, PALERMO
  - Divisione Di Ematologia, Ospedali Riuniti, Reggio Calabria, Reggio Calabria
  - Cattedra E Divisione Di Ematologia, Università Tor Vergata, Ospedale S.Eugenio, Roma, ROMA
  - Divisione Universitaria Ematologia - Az.Osp. San Giovanni Battista, Torino, TORINO
  - Ematologia, Azienda Ospedaliera S.Giovanni Battista, Torino, TORINO

REFERENCES:
- [Background] Buzaid AC, Durie BG. Management of refractory myeloma: a review. J Clin Oncol. 1988 May;6(5):889-905. doi: 10.1200/JCO.1988.6.5.889. PMID 2452861
- [Background] Palumbo A, Giaccone L, Bertola A, Pregno P, Bringhen S, Rus C, Triolo S, Gallo E, Pileri A, Boccadoro M. Low-dose thalidomide plus dexamethasone is an effective salvage therapy for advanced myeloma. Haematologica. 2001 Apr;86(4):399-403. PMID 11325646
- [Background] Palumbo A, Bringhen S, Bertola A, Cavallo F, Falco P, Massaia M, Bruno B, Rus C, Barbui A, Caravita T, Musto P, Pescosta N, Rossini F, Vignetti M, Boccadoro M. Multiple myeloma: comparison of two dose-intensive melphalan regimens (100 vs 200 mg/m(2)). Leukemia. 2004 Jan;18(1):133-8. doi: 10.1038/sj.leu.2403196. PMID 14586481
- [Background] Richardson PG, Barlogie B, Berenson J, Singhal S, Jagannath S, Irwin D, Rajkumar SV, Srkalovic G, Alsina M, Alexanian R, Siegel D, Orlowski RZ, Kuter D, Limentani SA, Lee S, Hideshima T, Esseltine DL, Kauffman M, Adams J, Schenkein DP, Anderson KC. A phase 2 study of bortezomib in relapsed, refractory myeloma. N Engl J Med. 2003 Jun 26;348(26):2609-17. doi: 10.1056/NEJMoa030288. PMID 12826635
- [Background] Barlogie B, Shaughnessy J, Tricot G, Jacobson J, Zangari M, Anaissie E, Walker R, Crowley J. Treatment of multiple myeloma. Blood. 2004 Jan 1;103(1):20-32. doi: 10.1182/blood-2003-04-1045. Epub 2003 Sep 11. PMID 12969978